CLINICAL TRIAL: NCT02565199
Title: Premotor Cortex: A New Target for Stroke Motor Rehabilitation Using Transcranial Magnetic Stimulation
Brief Title: Premotor Cortex: A New Target for Stroke Motor Rehabilitation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is temporarily suspended pending additional funding to continue subject recruitment.
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Cathrin Buetefisch, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00081901
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single motor training only (Experimental): For a pilot experiment, healthy, right-handed subjects will complete one testing session. During the testing session, subjects will complete motor training. The results of this experiment will determine the motor training protocol used in the main experiment.
  Interventions: Other: Motor Training
- Repetitive TMS during motor training (Experimental): Healthy, right-handed subjects will complete five testing sessions. During each testing session, subjects will complete motor training while receiving one of five repetitive transcranial magnetic stimulation (rTMS) protocols. Subjects will receive a different rTMS protocol at each testing session. By the end of the study, each subject will have received all rTMS protocols.
  Interventions: Device: rTMS over Premotor Cortex (Contralateral Hemisphere); Device: rTMS over Premotor Cortex (Ipsilateral Hemisphere); Device: rTMS (Control 1); Device: rTMS (Control 2); Device: rTMS (Control 3); Other: Motor Training

INTERVENTIONS:
Device: rTMS over Premotor Cortex (Contralateral Hemisphere) — * Location of rTMS: premotor cortex
  * Frequency of rTMS: 0.1 Hz
  * Time of rTMS: 50 milliseconds before the onset of movement-related EMG
  * Device: MagStim Super Rapid 2 Transcranial Magnetic Stimulator
  Arms: Repetitive TMS during motor training
Device: rTMS over Premotor Cortex (Ipsilateral Hemisphere) — * Location of rTMS: premotor cortex
  * Frequency of rTMS: 0.1 Hz
  * Time of rTMS: 50 milliseconds before the onset of movement-related EMG
  * Device: Super Rapid 2 Transcranial Magnetic Stimulator
  Arms: Repetitive TMS during motor training
Device: rTMS (Control 1) — * Location of rTMS: premotor cortex
  * Frequency of rTMS: 0.1 Hz
  * Time of rTMS: 400 milliseconds after the onset of movement-related EMG
  * Device: Super Rapid 2 Transcranial Magnetic Stimulator
  Arms: Repetitive TMS during motor training
Device: rTMS (Control 2) — * Location of rTMS: somatosensory cortex
  * Frequency of rTMS: 0.1 Hz
  * Time of rTMS: 50 milliseconds before the onset of movement-related EMG
  * Device: Super Rapid 2 Transcranial Magnetic Stimulator
  Arms: Repetitive TMS during motor training
Device: rTMS (Control 3) — * Location of rTMS: premotor cortex
  * Frequency of rTMS: 0.1 Hz
  * Time of rTMS: 50 milliseconds before the onset of movement-related EMG
  * Device: Super Rapid 2 Transcranial Magnetic Stimulator with Sham Coil
  Arms: Repetitive TMS during motor training
Other: Motor Training — During motor training, participants will quickly extend their hand at a pace of one extension every 5 seconds (0.2Hz) in response to an auditory cue.

SUMMARY:
The goal of the study is to determine the effect of repetitive transcranial magnetic stimulation (rTMS) over the premotor cortex on training-related improvements in motor performance and associated neural plasticity.

DETAILED DESCRIPTION:
Motor training is an important part of recovery after stroke. During motor training, stroke patients practice performing a movement and become better at performing the trained movement over time. Repetitive transcranial magnetic stimulation (rTMS), which uses magnetism to excite neurons near the surface of the brain, may further improve performance. Healthy adults made larger training-related improvements in their motor performance when they received rTMS over the primary motor cortex during motor training. There is evidence that the premotor cortex may be a more effective target than the primary motor cortex for rTMS for some stroke survivors. In the current study, the investigator will determine the effect of rTMS over the premotor cortex on training-related improvements in motor performance in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Motor training only (pilot participants):

* Have the ability to give informed, written consent
* Be aged 18-80 years old
* Be right-handed using the Edinburgh handedness inventory
* Have intact cognitive abilities (score higher than 75th percentile on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS))
* No current depression (score less than 7 on the Hamilton Depression Rating Scale (HDRS))
* No neurological disease
* No contradictions to Transcranial Magnetic Stimulation (TMS)
* TMS over the extensor carpi ulnaris (ECU) hotspot must evoke a motor evoked potential (MEP) in the ECU muscle
* MEP amplitude must increase by at least 20% as the TMS intensity increases
* The subjects must be comfortable when receiving TMS of all strengths.

Remaining study participants:

* Have the ability to give informed, written consent
* Be aged 55-80 years old
* Be right-handed using the Edinburgh handedness inventory
* Have intact cognitive abilities (score higher than 75th percentile on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS))
* No current depression (score less than a 7 on the Hamilton Depression Rating Scale (HDRS))
* No neurological disease
* No contradictions to Transcranial Magnetic Stimulation (TMS)
* TMS over the extensor carpi ulnaris (ECU) hotspot must be able to evoke a motor evoked potential (MEP) in the ECU muscle
* MEP amplitude must increase by at least 20% as the TMS intensity increases
* The subjects must be comfortable when receiving TMS of all strengths.

Exclusion Criteria:

* Impaired cognitive abilities (score lesser than 75th percentile on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS))
* Current depression (score more than 7 on the Hamilton Depression Rating Scale (HDRS))
* Neurological disease
* Has a contradiction to TMS
* MEP cannot be evoked with TMS in the ECU muscle
* Inability to tolerate one or more TMS strengths

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in wrist acceleration | Baseline, post-motor training (1 minute, 30 minutes and 60 minutes after completion of motor training)
  The subjects will be asked to perform 7 isometric wrist extensions before and after motor training. Wrist acceleration will be measured by a gyroscope taped to the dorsum of the subject's hand undergoing motor training. An increase in the maximum acceleration that persists at least an hour after training is indicative of motor learning. We will compare the effect of the rTMS protocols on the change in the wrist acceleration associated with motor learning (baseline to post 1 min, baseline to post 30 mins, baseline to post 60 mins).
Change in stimulus response curve (SRC) | Baseline, post-motor training (1 minute, 30 minutes and 60 minutes after completion of motor training)
  The stimulus response curve (SRC) is a set of motor evoked potentials (MEPs) collected in response to transcranial magnetic stimulation (TMS) pulses of increasing intensities. The SRC can characterize input-output parameters of the corticospinal tract and organization of the primary motor cortex. A change in the SRC parameters after training will reflect a change in the organization of the primary motor cortex associated with motor learning. We will compare the effect of the rTMS protocols on the change in the SRC parameters associated with motor learning (baseline to post 1 min, baseline to post 30 mins, baseline to post 60 mins).
Change in short interval intracortical inhibition (SICI) | Baseline, post-motor training (1 minute, 30 minutes and 60 minutes after completion of motor training)
  Short interval intracortical inhibition (SICI) is an inhibitory phenomenon in the motor cortex. To test for SICI, a sub-threshold conditioning stimulus (CS) will precede a supra-threshold test stimulus (TS) by 2 milliseconds (ms). The amplitude of a conditioned TS-evoked MEP will be expressed as a percent of the amplitude of an unconditioned TS-evoked MEP. A decrease in the percent MEP after training would indicate a increase in SICI. An increase in the percent MEP after training would indicate a decrease in SICI. We will compare the effect of the rTMS protocols on the change in SICI associated with motor learning (baseline to post 1 min, baseline to post 30 mins, baseline to post 60 mins).

SECONDARY OUTCOMES:
Change in wrist force | Baseline, post-motor training (1 minute, 30 minutes and 60 minutes after completion of motor training)
  The subjects will be asked to perform 7 isometric wrist extensions before and after motor training. A force transducer transducer will record the maximum force produced during the wrist extensions.
Change in reaction time | Baseline and post-motor training (1 minute, 30 minutes and 60 minutes after completion of motor training)
  Subjects will be asked to perform 7 auditory-cued ballistic wrist extensions before and after motor training. Electomyographic (EMG) activity recorded during the ballistic wrist extensions will be used to measure reaction time. Reaction time is the length of time between the auditory cue and the onset of the movement-related EMG burst of the extensor carpi ulnaris (ECU) muscle.
Change in task accuracy | Baseline and post-motor training (1 minute after completion of motor training)
  Task accuracy will be determined by the number of successful trials over the number of total trials. A trial will be considered successful when the subject moves a cursor from the home position into a target box by modulating the acceleration of their wrist. An increase in task accuracy after training will indicate motor learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States